CLINICAL TRIAL: NCT05210673
Title: Enhanced Recovery for Patients Undergoing Radical Cystectomy. A Randomized Controlled Study
Brief Title: Enhanced Recovery for Patients Undergoing Radical Cystectomy.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menoufia University (Other)
Collaborators: Ezzeldin Saleh Ibrahim (Unknown); asmaa mohamed hamza (Unknown); asmaa ibrahim mohamed (Unknown); mohamed marzouk abdallah (Unknown)
Responsible Party: Principal Investigator, ashraf magdy eskandr, assistant professor of anesthesia, Menoufia University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: ERAS in radical cystectomy
Record Dates: First submitted 2022-01-14; First posted 2022-01-27 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-01

CONDITIONS: Post Procedural Discharge

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group A (Experimental): non ERAS pathway
  Interventions: Other: Non ERAS pathway
- group B (Active Comparator): ERAS pathway
  Interventions: Other: ERAS

INTERVENTIONS:
Other: ERAS — Preoperative: Preoperative explanation of ERAS. Preoperative medical optimization. Smoking cessation 4-8 weeks before surgery. Nutritional status assessment. Preoperative fasting: 2hours for Clear fluids and water, 6hours for Semi-solid foods and 8 hours for Solid food. Preoperative carbohydrate loading. Pre-anesthetic medication: Avoid long active sedatives. Thromboembolic prophylaxis and Compression stockings Intraoperative: Antimicrobial prophylaxis and skin preparation. Epidural analgesia. Prevention of intraoperative hypothermia. Intraoperative fluid management. Minimize incision. Drain strategy Postoperative: Nasogastric intubation. Early oral intake. Early mobilization. Prevention of postoperative ileus through. Prevention of postoperative nausea and vomiting. Multimodal opioid sparing analgesia. Discharge criteria: Patients have resumed adequate oral intake and normal bowel function, Effective oral pain management and No other clinical or biochemical concerns
  Arms: group B
Other: Non ERAS pathway — standard preoperative preparation intraoperative: combined general and epidural anesthesia postoperative standard care
  Arms: group A

SUMMARY:
Investigators hypothesize that with the use of enhanced recovery of surgery (ERAS), the postoperative hospital stay after radical cystectomy is reduced, and also postoperative complications are decreased.

DETAILED DESCRIPTION:
Radical cystectomy (RC) is believed to be associated with high morbidity and prolonged length of hospital stay even with advances in perioperative medical care. Enhanced Recovery After Surgery (ERAS) pathways are multidisciplinary, multimodal evidence-based approaches to perioperative protocol by which patients are treated. The most important aims of this multimodal approach are modifying as many of the factors contributing to the morbidity of RC as possible, the improvement of patients' preoperative status, and the perioperative maintenance of homeostasis by minimizing stress response and inflammation to improve patient outcomes and decrease the length of inpatient hospital stay. The investigators hypothesize that with the use of enhanced recovery of surgery (ERAS), the postoperative hospital stay after radical cystectomy is reduced, and also postoperative complications are decreased.

ELIGIBILITY:
Inclusion Criteria:

* Age: 40-85 years.
* Adequate cognitive state (able to understand and collaborate)
* American society of anesthesia (ASA) I, II and III.

Exclusion Criteria:

* ASA IV

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
length of hospital stay | 1-15 days
  length of hospital stay in days

SECONDARY OUTCOMES:
Onset of bowel movement | 1-5 days
  Onset of bowel movement in days
Onset of early mobilization | 1-15 days
  Onset of early mobilization in days
Postoperative analegesic consumption | 1-15 days
  opioid and paracetamol

CONTACTS AND LOCATIONS:
Overall Officials: ashraf M eskandr, Study Director — menoufia faculty of medicine
Locations (1):
- Ashraf Magdy Eskandr, Shibeen Elkoom, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
when requested from authors